CLINICAL TRIAL: NCT00888810
Title: A Phase II Study Evaluating the Association of Topotecan and Lapatinib in Early Recurrent (Less Than 12 Months)Ovarian or Peritoneal Cancer Patients After First Line of Platinum-Based Chemotherapy
Brief Title: Efficacy of Topotecan and Lapatinib in Early Recurrent Ovarian or Peritoneal Cancer
Acronym: TOPO-LAPA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of efficacy (intermediate analysis)
Sponsor: Centre Francois Baclesse (Other)
Collaborators: GlaxoSmithKline (Industry); Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Pr Florence JOLY - MD-PHD, Centre François Baclesse
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-005706-44
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Cancer; Ovarian; Relapse; Chemotherapy
Keywords: ovarian - cancer - relapse - topotecan - lapatinib
MeSH Terms: conditions — Neoplasms; Recurrence | interventions — Topotecan; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: TOPOTECAN — IV administration on Day 1, day 8 and day 15, at the dose level of 3.2 mg/m² for 6 cycles of 28 days(up to 8 cycles)
  Other Names: HYCAMTIN
Drug: LAPATINIB — Daily oral administration during all the study. 1250 mg/day
  Other Names: TYVERB

SUMMARY:
The objective of the trial was to evaluate the efficacy of the association of topotecan and lapatinib in patients who failed first line platinum-based chemotherapy within 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age superior or equal 18 years
* primitive ovarian adenocarcinoma histologically confirmed
* or peritoneal or fallopian tube adenocarcinoma histologically confirmed
* Progression or relapse within 12 months after the end of first line of platin based chemotherapy
* association in first line with other anticancer agent is allowed (taxanes, anthracyclines, alkylants or gemcitabine) and with an anti-angiogenic (bevacizumab, sunitinib).
* intra-peritoneal chemotherapy in first line is possible
* No previous treatment with HER inhibitors (ex : gefitinib)
* HER status not necessary
* measurable lesions (RECIST criteria). and/or CA125 value higher than 2 fold the normal value or CA125 higher than 2 fold nadir value (if no normalized) proved by two samples distant of 1 month
* OMS inferior or equal 2.
* biological parameters as follow: creatininemia ≤ 150 µmol/L or clearance ≥ 50 mL/min,bilirubin ≤ 1,5 LNS,transaminases and or alcalin phosphatases ≤ 2 LNS without hepatic metastasis or ≤ 3 LNS if hepatic metastasis,neutrophils ≥ 1,5.109/L,plaquettes ≥ 100.109/L.
* normal FEV
* No previous treatment by chemotherapy, hormonotherapy, immunotherapy or radiotherapy within 4 weeks before inclusion
* No concomitant treatment forbidden with lapatinib.
* No previous treatment by Amiodarone in 6 months before inclusion
* signed informed consent

Exclusion Criteria:

* Previous treatment with :

  * intensive chemotherapy with autograft
  * two lignes of chemotherapy
  * previous total abdominal irradiation
  * previous chemotherapy with anti-HER treatment
* History of brain or meningitis metastasis uncontrolled.
* Malignancies except for adequately treated carcinoma in situ of the cervix and/or basal cell skin cancer.
* uncontrolled infectious pathology
* uncontrolled cardiovascular disease
* Patients with an active intestinal occlusion not permit oral treatment
* known hypersensibility to topotecan and its excipients
* Woman of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period
* Individual deprived of liberty

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-03

PRIMARY OUTCOMES:
Evaluation of global response rate (complete response, partial response and stable disease)of the association topotecan-lapatinib. | every two cycles of chemotherapy

SECONDARY OUTCOMES:
Global survival rate, survival rate without progression, response time, time without progression, safety, quality of life, Caracterisation of biological response (tumor, ascite and blood samples) | each cycle of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Florence JOLY, MD-PHD, Principal Investigator — Centre François Baclesse
Locations (21):
- France (21):
  - Centre François Baclesse, Caen, CALVADOS
  - Centre Paul Papin, Angers
  - CHU Jean MINJOZ, Besançon
  - Institut Bergonié, Bordeaux
  - Centre G-F Leclerc, Dijon
  - CHD Les Oudairies, La Roche-sur-Yon
  - Centre Jean Bernard, Le Mans
  - Centre Val d'Aurelle, Montpellier
  - Centre azuréen de cancérologie, Mougins
  - Centre Alexis vautrin, Nancy
  - Centre Catherine de Sienne, Nantes
  - Centre René Gauducheau, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hôpital Diaconesses, Paris
  - Institut CURIE, Paris
  - APHP Hopital TENON, Paris
  - Institut Jean Godinot, Reims
  - Institut de Cancérologie de la Loire, Saint-Etienne
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- See also: French National Protocol Registration System — http://www.e-cancer.fr